CLINICAL TRIAL: NCT06950099
Title: Pathophysiological Evaluation of Idiopathic Intracranial Hypertension Using Glymphatic and Connectomic Imaging
Brief Title: Advanced Neuroimaging in Idiopathic Intracranial Hypertension
Acronym: IIH
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: American Headache Society (Other)
Responsible Party: Sponsor
Other Study IDs: JT44344 fMRI in IIH
Record Dates: First submitted 2025-03-24; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Intracranial Hypertension (IIH); Glymphatic System
Keywords: idiopathic intracranial hypertension; MRI; diffusion tensor imaging; IIH
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with TSS: Pre- and post-stenting

SUMMARY:
Idiopathic intracranial hypertension (IIH) is characterized by elevated intracranial pressure leading to symptoms like papilledema, headache, and cognitive dysfunction. While the etiology is complex, abnormal cerebrospinal fluid dynamics due to venous outflow restriction from transverse sinus stenosis (TSS) is common. TSS may disrupt the glymphatic system, a brain-wide network facilitating cerebrospinal fluid and interstitial fluid exchange, by impairing CSF absorption, altering perivascular space dynamics, and disrupting pressure gradients crucial for waste clearance. Venous sinus stenting (VSS) can improve symptoms in many patients by alleviating venous congestion, but its effects on glymphatic function are unclear. This prospective study aims to evaluate novel quantitative brain imaging metrics as surrogate markers to better understand IIH pathophysiology before and after VSS in patients with refractory IIH and TSS. The investigators will use advanced MRI techniques, including MR elastography (MRE) to assess brain stiffness, diffusion tensor imaging (DTI) to evaluate water diffusion, arterial spin labeling (ASL) imaging to measure blood-brain barrier (BBB) permeability, and functional MRI to analyze pain networks. The investigators hypothesize that 1) these noninvasive imaging metrics will correlate with the degree of venous congestion and changes after venous sinus stenting (VSS) and 2) the imaging findings will correlate with clinical treatment outcomes. By correlating imaging markers with venous pressures and symptom changes, the investigators aim to gain insights into IIH mechanisms, expand diagnostic tools, and potentially guide clinical decision-making and treatment response monitoring. The overarching goal is to better understand IIH's underlying pathophysiology, which could lead to improved diagnostic criteria, more targeted treatments, and better prediction of treatment outcomes for patients with this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

• Refractory IIH patients who require and plan to have a venous sinus stenting

Exclusion Criteria:

* History of head trauma and shunting or leak repair
* Major concurrent, active non-cephalic pain syndrome
* Contradictions for MRIs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Refractory IIH patients who require and plan to have a venous sinus stenting
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Advanced MRI measurements changes pre- and post-stenting | 3 months
  DTI-ALPS index

SECONDARY OUTCOMES:
Clinical headache outcomes | 3 months
  Monthly headache days

OTHER OUTCOMES:
Questionnaire outcomes | 3 months
  Quality of life using Physicians Global Assessment (from 0 to 10, 0=free of complaints, 10=strong discomfort),

CONTACTS AND LOCATIONS:
Overall Officials: Hsiangkuo Yuan, MD PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided